CLINICAL TRIAL: NCT03196765
Title: Phase I/II, Open-Label, Dose Escalation Study of the Safety, Pharmacokinetics and Pharmacodynamics of NV1205 in Pediatric Male Subjects With Childhood Cerebral Adrenoleukodystrophy (CCALD)
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of NV1205 in Pediatric Male Subjects With Adrenoleukodystrophy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: NeuroVia, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NV1205-009
Record Dates: First submitted 2017-05-05; First posted 2017-06-23 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-05

CONDITIONS: X-Linked Adrenoleukodystrophy
Keywords: X-ALD
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — GC 1 compound

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sobetirome (NV1205) — Once a day oral dose of the study drug
  Other Names: NV1205

SUMMARY:
This is a phase I/II, open label dose escalation study of multiple dose levels of NV1205 with a long-term treatment phase.

DETAILED DESCRIPTION:
This study is to evaluate the safety, pharmacokinetics, and efficacy of NV1205 in pediatric patients diagnosed with childhood cerebral adrenoleukodystrophy (CCALD).

The study consists of:

* Screening period: within 30 days of first dose
* Main treatment period of 12 weeks (Part 1- from Screening to Week 12)
* Long Term Treatment (LTT) period (Part 2- Week 13 through Week 96)

In Part 1, subjects will have an initial 4-week treatment period at the assigned dose and, if no safety concerns are noted, subjects continue for another 8 weeks of extended safety assessment.

There will be several cohorts of subjects enrolled. After each Cohort has completed the 4-week initial safety assessment, the safety data will be reviewed by an independent Data Safety Monitoring Board (DSMB) and, subject to DSMB recommendation, Cohort 2 will be enrolled and receive the next dose level. After Cohort 2 has completed 4 weeks of treatment, the DSMB will review all available safety data (Cohorts 1 and 2) and, subject to DSMB recommendation, Cohort 3 will be enrolled and receive the next dose level. Additional Cohorts may be enrolled at the recommendation of the DSMB with an incremental dose increase.

In Part 2, subjects will continue to receive treatment in the LTT period of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥4 years and <18 years of age
2. CCALD diagnosis confirmed by genetic testing
3. Loes score of >0 and ≤15
4. Patients on VLCFA lowering agents such as Lorenzo's oil must stop the medication and have high VLCFA levels before enrollment

Exclusion Criteria:

* Significant medical conditions such as heart, thyroid, or liver disease
* HSCT recipients

Ages: 4 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Adverse events

SECONDARY OUTCOMES:
Area under the curve concentration of NV1205 in plasma | 12 weeks
  A sparse sampling approach will be utilized to estimate a 24-hr area under the curve of NV1205 plasma concentration

OTHER OUTCOMES:
Loes score | 2 years
  Percent change from baseline in brain lesions assessed as Loes score will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: John Henderson, MD, Study Director — NeuroVia, Inc.
Locations (13):
- Argentina (2):
  - Hospital Austral, Buenos Aires
  - Hospital General de ninos Pedro de Elizalde, Buenos Aires
- Monash Health, Clayton, Victoria, Australia
- Chile (2):
  - Hospital Clínico San Borja Arriarán, Santiago
  - Hospital Dr. Luis Calvo Mackenna, Santiago
- Fundacion Cardioinfantil, Bogotá, Colombia
- Hôpital Bicêtre - Paris Sud, Paris, France
- Russia (3):
  - Endocrinology Research Center, Moscow
  - Moscow Morozov's Children Clinical Hospital, Moscow
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg
- National Children's Specialized Hospital 'OKHMATDET', Kiev, Ukraine
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No